CLINICAL TRIAL: NCT01954784
Title: A Study of Low-dose Lenalidomide After Non-myeloablative Allogeneic Stem Cell Transplant With Bortezomib as GVHD Prophylaxis in High Risk Multiple Myeloma
Brief Title: Lenalidomide After Donor Stem Cell Transplant and Bortezomib in Treating Patients With High Risk Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1A13; NCI-2013-01777 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE1A13 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — fludarabine phosphate; Whole-Body Irradiation; Cyclosporine; Mycophenolic Acid; Bortezomib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nonmyeloablative alloHSCT, lenalidomide) (Experimental): PREPARATIVE REGIMEN: Patients receive fludarabine phosphate on days -5 to -3 and undergo TBI on day -1.
  TRANSPLANT: Patients undergo allogeneic hematopoietic SCT on day 0.
  GVHD PROPHYLAXIS: Patients receive standard GVHD prophylaxis comprising cyclosporine PO BID beginning on day -1 with taper beginning on day 100, mycophenolate mofetil PO BID on days 1-56, and bortezomib SC weekly from day 1 to day 91.
  MAINTENANCE THERAPY: Beginning on day 100, patients receive lenalidomide PO daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fludarabine phosphate; Radiation: total-body irradiation; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Drug: cyclosporine; Drug: mycophenolate mofetil; Drug: bortezomib; Drug: lenalidomide; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: fludarabine phosphate
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — Undergo nonmyeloablative allogeneic hematopoietic SCT
Drug: cyclosporine — Given PO
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given PO
  Other Names: Cellcept; MMF
Drug: bortezomib — Given SC
  Other Names: LDP 341; MLN341; VELCADE
Drug: lenalidomide — Given PO
  Other Names: CC-5013; IMiD-1; Revlimid
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of lenalidomide after donor stem cell transplant and bortezomib in treating patients with high-risk multiple myeloma. Giving low doses of chemotherapy and total-body irradiation before a donor stem cell transplant helps stop the growth of cancer cells. It may also the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving a bortezomib at the time of transplant may stop this from happening. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Giving lenalidomide after donor stem cell transplant may be an effective treatment for multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify the maximal tolerated dose (MTD) and safety of lenalidomide up to 10mg following non-myeloablative allogeneic stem cell transplant for multiple myeloma.

SECONDARY OBJECTIVES:

I. Assess safety and tolerability of weekly bortezomib following non-myeloablative allogeneic stem cell transplant.

II. Obtain estimates of non-relapse mortality. III. Obtain estimates of acute and chronic graft-versus-host disease (GVHD). IV. Obtain estimates of 1 year relapse and survival.

OUTLINE: This is a dose-escalation study of lenalidomide.

PREPARATIVE REGIMEN: Patients receive fludarabine phosphate on days -5 to -3 and undergo total body irradiation (TBI) on day -1.

TRANSPLANT: Patients undergo allogeneic hematopoietic stem cell transplant (SCT) on day 0.

GVHD PROPHYLAXIS: Patients receive standard GVHD prophylaxis comprising cyclosporine orally (PO) twice daily (BID) beginning on day -1 with taper beginning on day 100, mycophenolate mofetil PO BID on days 1-56, and bortezomib subcutaneously (SC) weekly from day 1 to day 91.

MAINTENANCE THERAPY: Beginning on day 100, patients receive lenalidomide PO daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up monthly for 1 year post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic multiple myeloma by International Myeloma Working Group (IMWG) criteria according to the most recent updated version (International Myeloma Workshop [IMW] meeting in Paris 2011)
* Must have received at least 3 of the following classes of anti-myeloma agents either alone or in combination: glucocorticoids, immunomodulatory drugs including thalidomide, proteasome inhibitors, alkylating chemotherapy, or anthracyclines
* Must meet any of these criteria for high risk disease:

  * Relapse or progressive disease according to uniform response criteria within 2 years after starting first-line therapy or within 2 years after autologous stem cell transplant
  * Failure to achieve partial response (PR) within 6 months of staring first-line therapy
  * Presence of high risk cytogenetic features (t(14;16), t(14;20), deletion 17p)
  * Chromosome 14 translocations other than to chromosome 11
  * Chromosome 1p deletion and 1q amplification
  * MyPRS gene expression score equal or higher than 45.2
  * High risk 70 gene expression profile (MyPRS GEP70TM)
  * Any other high risk genetic profile that is determined by future IMWG consensus or by internal myeloma panel consensus; for the latter, any additional criteria will be submitted as an addendum
  * Diagnosis with multiple myeloma between the ages of 18-50
* Must have achieved at least a minor response to any previous regimen according to adapted European Group for Blood and Marrow Transplantation (EBMT) criteria
* Must have suitable matched sibling or matched unrelated donor for stem cell source
* Must be transplant-eligible per institution guidelines
* Must have estimated glomerular filtration rate (eGFR) by Modification of Diet in Renal Disease (MDRD) formula or Cockroft-Gault formula of 50mL/min or higher
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of Revlimid REMS®
* Females of childbearing potential must have negative serum or urine pregnancy test and use acceptable birth control methods
* Able to take aspirin daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid [ASA] may use warfarin or low molecular weight heparin)

Exclusion Criteria:

Participants must not:

* Have known hypersensitivity to thalidomide or lenalidomide
* Have progressive disease at the time of transplant
* Uncontrolled concurrent significant medical or psychological co-morbidity
* Grade 3 peripheral neuropathy
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV); patients who are seropositive because of hepatitis B virus vaccine are eligible
* Be females who are pregnant
* Recent (within 3 years) history of other malignancies, excluding basal cell carcinoma or squamous cell carcinoma of the skin
* Be currently enrolled in another investigational treatment protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-10-07 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
MTD of lenalidomide defined as one dose level below the dose in which 2 or more patients at a specified dose level experience dose limiting toxicity (DLT) according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (v. 4.0) | Day 128 post-transplant

SECONDARY OUTCOMES:
Safety assessed by evaluating the incidence of toxicity according to CTCAE v. 4.0 | Up to day 100
Incidence of acute GVHD according to Center for International Blood and Marrow Transplant Research (CIBMTR) | 1 year
Incidence of chronic GVHD according to National Institutes of Health (NIH) | 1 year
Time to deaths without relapse/recurrence | 1 year
Progression-free survival | From study entry to progression as defined by international response criteria or death of any cause, whichever comes first, assessed at 1 year
Overall survival | From study entry to death from any cause, assessed at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hien K Liu, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States